CLINICAL TRIAL: NCT02782923
Title: Driving After Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-01224
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Cervical Disc Disease
Keywords: Cervical Spine Surgery; Simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- s-ACDFwith STISIM (Experimental): Single-level anterior cervical discectomy fusion
  Interventions: Device: STISIM driving simulator
- m-ACDF with STISIM (Experimental): Multi-level anterior cervical discectomy and fusion
  Interventions: Device: STISIM driving simulator
- CDR with STISIM (Experimental): Cervical disc replacement
  Interventions: Device: STISIM driving simulator
- PCLF with STISIM (Experimental): Posterior laminectomy and fusion
  Interventions: Device: STISIM driving simulator
- PCD with STISIM (Experimental): Posterior cervical decompression procedure
  Interventions: Device: STISIM driving simulator
- Control Group with STISIM (Sham Comparator)
  Interventions: Device: STISIM driving simulator

INTERVENTIONS:
Device: STISIM driving simulator — This simulator is complete with computerized driving scenarios and driving hardware, has been validated in numerous studies and allows for a more comprehensive investigation of driving performance. The simulated course recreates standard turns, traffic intersections, pedestrian crosswalks, lane changes and several hazardous conditions routinely encountered during driving situations.

SUMMARY:
This is a single-center, prospective controlled simulation study designed comparing and evaluating the driving performance of subjects who have had cervical spine surgery and the use of a validated driving simulator. To date, there haven't been evidence-based recommendations to determine a patient's "fitness to drive" in the peri-operative or postoperative state. The objective of this study is to delineate the effect cervical spine procedures have on driving performance in the peri-operative time period. The study will take place at New York University Langone Medical Center - Hospital for Joint Diseases which will include the surgeries. The follow up visits will be at the NYU Center for Musculoskeletal Care.

ELIGIBILITY:
Inclusion Criteria:

Study Subjects

* Age between 18 and 80 years
* Indicated for elective cervical spine surgery (including ACDF [single or multilevel], posterior cervical laminectomy and fusion, posterior cervical laminoplasty, posterior cervical foraminotomy, cervical disc replacement) after failing at least 6 weeks of non-operative treatment modalities
* Valid driving license
* Regular use of a vehicle
* Signed consent form

Inclusion Criteria

Control Subjects:

* Age between 18 and 80 years
* No pre-existing or recent injuries to neck, torso, back
* No neurologic or systemic debilitating conditions
* Valid driving license
* Regular use of a vehicle
* Signed consent form

Exclusion Criteria:

* Significant visual impairment
* Significant debilitating neurological condition with loss of function of one or more extremities
* Recent extremity surgery
* Recent eye surgery
* Previous history of motion sickness, vertigo in simulated settings
* Recent history of chemical or narcotic dependency involved in active litigation related to their spine problem a the time of screening.
* Involved in workers compensation related to their spine problem at the time of screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-12; Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Kim, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical Surgical Patients: Participants who have undergone cervical spine surgery
Period: Overall Study
Arm/Group | Cervical Surgical Patients
Started | 19
Completed | 4
Not Completed | 15
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Arm/Group | Cervical Surgical Patients
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 47 [30 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Total Collisions (TC)
Description: Change from Baseline in Overall collisions (BL-3mo). Includes both "off-road" and "on-road" collisions.
Time Frame: Baseline, 3 months
Measure: Median (Full Range); unit: collisions/crashes
Arm/Group | Cervical Surgical Patients
Number analyzed (Participants) | 4
collisions/crashes | 2 [0 to 4]

2. Primary Outcome: Change in Number of Centerline Crossings (CC)
Description: Change from baseline in the number of unsafe lane changes. Measured by the number of times the patient failed to check blind spots when changing lanes or changed lanes when another "vehicle" was in the patient's blind spot.
Time Frame: Baseline, 3 months
Measure: Median (Full Range); unit: centerline crossings
Arm/Group | Cervical Surgical Patients
Number analyzed (Participants) | 4
centerline crossings | 1.5 [0 to 2]

3. Primary Outcome: Change in Number of Off-road Excursions (ORE)
Description: Number of off-road excursions was measured by the number of times the patient's "vehicle" traversed the lateral road edge and traveled off onto the grass
Time Frame: Baseline, 3 months
Measure: Median (Full Range); unit: off-road excursions
Arm/Group | Cervical Surgical Patients
Number analyzed (Participants) | 4
off-road excursions | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cervical Surgical Patients
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT02782923/Prot_000.pdf